CLINICAL TRIAL: NCT00541385
Title: Phase III Comparative, Open-labelled, Randomised, Clinical Study to Assess a Fixed Dose of Oral Pyronaridine Artesunate Granule Formulation vs. Coartem® Crushed Tablets in Infants With Acute Uncomplicated Plasmodium Falciparum Malaria
Brief Title: Pyronaridine Artesunate 3:1 Granule Formulation vs. Coartem© Crushed Tablets in P. Falciparum Malaria Pediatric Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Shin Poong Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SP-C-007-07
Record Dates: First submitted 2007-10-09; First posted 2007-10-10 (Estimated); Results first posted 2021-11-22 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-10

CONDITIONS: Malaria
Keywords: Falciparum malaria; pediatric; Coartem; artesunate; lumefantrine; pyronaridine; Pyramax
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — pyronaridine tetraphosphate, artesunate drug combination; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PA group (Experimental): Oral pyronaridine/artesunate (PA, 60:20mg granules) once a day for 3 consecutive days (Days 0, 1, and 2).
  Posology based on body weight ranges.
  Interventions: Drug: pyronaridine artesunate
- AL group (Active Comparator): Oral artemether/lumefantrine (AL, 20:120mg crushed tablets) twice a day for 3 consecutive days (Days 0, 1, and 2).
  Posology based on body weight ranges.
  Interventions: Drug: arthemeter lumefantrine

INTERVENTIONS:
Drug: pyronaridine artesunate — The strength of the granule formulation is 60:20 mg pyronaridine artesunate per sachet. Depending on their body weight, patients will receive between 1 to 3 pyronaridine artesunate sachets per day, for 3 consecutive days The actual dose-range covered by this regimen is 7.0:2.3 mg/kg to 13.3:4.4 mg/kg pyronaridine artesunate, which has shown to be effective and safe in the phase II studies conducted in children and adults.
  Other Names: Pyramax
  Arms: PA group
Drug: arthemeter lumefantrine — The strength of the tablet is 20 mg artemether and 120 mg lumefantrine. Depending on their body weight, patients will receive either 1 or 2 crushed tablets twice a day (≥5 to <15 = 1 tablet, 15 to <25 kg = 2 tablets), for 3 consecutive days.
  Other Names: Coartem
  Arms: AL group

SUMMARY:
The primary objective of this Phase III clinical study is to demonstrate the efficacy of the fixed combination of pyronaridine artesunate (PA) granule formulation (60:20 mg; pediatric PYRAMAX®) by showing a PCR-corrected adequate clinical and parasitological cure rate (ACPR) of more than 90%.

Secondary objectives of this clinical study are to compare the efficacy (non-inferiority) and safety of the PA granule formulation compared to Coartem® (ie, the combination of artemether/lumefantrine [AL]) crushed tablets in a paediatric population and to assess the safety of the PA granule formulation.

DETAILED DESCRIPTION:
This is a multi-centre, comparative, randomised, open-label, parallel-group study of the efficacy and safety of a 3-day regimen of a fixed combination of PA (3:1) versus AL in the treatment of acute uncomplicated Plasmodium falciparum mono-infection. The study population will include 534 patients, comprising male and female infants and children (body weight ≥5 and <25 kg) recruited from study sites in East, Central, and West Africa and South East Asia (max. 150 patients/site).

Patients will be randomised in a 2:1 ratio to receive either oral PA (60:20 mg granules) once a day for 3 consecutive days (Days 0, 1, and 2) or AL (20:120 mg crushed tablets) twice a day for 3 consecutive days (Days 0, 1, and 2). The study drug will be administered by a Third Party Investigator unblinded to the study treatment, while the Investigator will remain blinded. For PA, the dose range covered by this regimen is 7.0:2.3 mg to 13.3:4.4 mg, which has been shown to be effective and safe in Phase I and II studies. Posology will be based on body weight ranges for both the PA and AL regimens.

Patients will be confined to the study facility ≥4 days (Days 0, 1, 2, and 3) and remain near the study site for ≥7 days, or once fever and parasite clearance has been confirmed for ≥24 hours - whichever occurs earlier.

The primary efficacy end point for this study is the proportion of subjects with PCR-corrected ACPR on Day 28. Scheduled follow-up visits will continue until completion of the study at Day 42. In the case of adverse events reported and unresolved at Day 42, patients will be followed up for a further 30 days, or until resolution of the event.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≤12 years of age.
2. Body weight ≥ 5 kg and < 25 kg with no clinical evidence of severe malnutrition (defined as a child whose weight-for-height is below -3 standard deviations or <70% of the median of the NCHS/WHO normalised reference values).
3. Presence of acute uncomplicated P. falciparum mono-infection confirmed by:

   1. Fever, as defined by axillary temperature ≥37.5°C or oral/tympanic/rectal temperature ≥38°C, or documented history of fever in the previous 24 hours and,
   2. Positive microscopy of P. falciparum with parasite density between 1,000 and 200,000 asexual parasite count/µl of blood.
4. Written informed consent, in accordance with local practice, provided by parent/guardian. If the parent/guardian is unable to write, witnessed consent is permitted according to local ethical considerations. Where possible, patient assent will be sought.
5. Ability to swallow whole volume of liquid in which medication is suspended.
6. Female patients of child-bearing potential must be neither pregnant (as demonstrated by a negative pregnancy test) nor lactating, and must be willing to take measures to not become pregnant during the study period.
7. Ability and willingness to participate based on information given to parent or guardian and access to health facility. The patient is to comply with all scheduled follow up visits until D42.

Exclusion Criteria:

1. Patients with signs and symptoms of severe/complicated malaria requiring parenteral treatment according to the World Health Organization Criteria 2000 [Attachment 3].
2. Mixed Plasmodium infection.
3. Severe vomiting, defined as >3 times in the 24 hours prior to inclusion in the study or inability to tolerate oral treatment, or severe diarrhoea defined as ≥3 watery stools per day.
4. Known history or evidence of clinically significant disorders such as cardiovascular (including arrhythmia, QTc interval ≥450 milliseconds), respiratory (including active tuberculosis), history of jaundice, hepatic, renal, gastrointestinal, immunological (including active HIV-AIDS), neurological (including auditory), endocrine, infectious, malignancy, psychiatric, history of convulsions or other abnormality (including recent head trauma).
5. Presence of significant anaemia, as defined by Hb <8 g/dL.
6. Presence of febrile conditions caused by diseases other than malaria.
7. Known history of hypersensitivity, allergic or adverse reactions to pyronaridine, lumefantrine or artesunate or other artemisinins.
8. Patients with known disturbances of electrolytes balance, e.g. hypokalaemia or hypomagnesaemia.
9. Use of any other antimalarial agent within 2 weeks prior to start of the study as evidenced by reported patient history.
10. Pregnant or breastfeeding.
11. Patients taking any drug which is metabolised by the cytochrome enzyme CYP2D6 (flecainide, metoprol, imipramine, amitriptyline, clomipramine).
12. Received an investigational drug within the past 4 weeks.
13. Known active Hepatitis A IgM (HAV-IgM), Hepatitis B surface antigen (HBsAg) or Hepatitis C antibody (HCV Ab).
14. Known positive for HIV antibody.
15. Liver function tests [ASAT/ALAT levels] >2.5 times upper limit of normal range.
16. Known significant renal impairment as indicated by serum creatinine of >1.4 mg/dL.
17. Previous participation in any clinical study with pyronaridine artesunate.

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 535 (Actual)
Dates: Start 2007-10; Primary Completion 2008-09 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claude Oeuvray, PhD, Study Director — Medicines for Malaria Venture
Locations (8):
- Centre National de Recherche et de Formation sur le Paludisme, Ouagadougou, Burkina Faso
- Unité de Paludologie de l'Institut Pasteur d'Abidjan, Abidjan, Côte d’Ivoire
- Ecole de Santé Publique, Faculté de Médecine, Université de Kinshasa, Kinshasa, Democratic Republic of the Congo
- Medical Research Unit, Albert Schweitzer Hospital, Lambaréné, Gabon
- Siaya District Hospital, Medical Superintendent's office, Siaya, Kenya
- Malaria Research and Training Center, Faculté de Médecine, de Pharmacie et d'Ondonto-stomatologie, Bamako, Mali
- Instituto Nacional de Saude, Ministero de Saude, Maputo, Mozambique
- Puerto Princesa General Hospital, Puerto Princesa City, Philippines

REFERENCES:
- [Result] Kayentao K, Doumbo OK, Penali LK, Offianan AT, Bhatt KM, Kimani J, Tshefu AK, Kokolomami JH, Ramharter M, de Salazar PM, Tiono AB, Ouedraogo A, Bustos MD, Quicho F, Borghini-Fuhrer I, Duparc S, Shin CS, Fleckenstein L. Pyronaridine-artesunate granules versus artemether-lumefantrine crushed tablets in children with Plasmodium falciparum malaria: a randomized controlled trial. Malar J. 2012 Oct 31;11:364. doi: 10.1186/1475-2875-11-364. PMID 23113947
- [Derived] Ramharter M, Djimde AA, Borghini-Fuhrer I, Miller R, Shin J, Aspinall A, Richardson N, Wibberg M, Fleckenstein L, Arbe-Barnes S, Duparc S. Safety and efficacy of pyronaridine-artesunate paediatric granules in the treatment of uncomplicated malaria in children: insights from randomized clinical trials and a real-world study. Malar J. 2024 Feb 28;23(1):61. doi: 10.1186/s12936-024-04885-3. PMID 38418982
- [Derived] Ayyoub A, Methaneethorn J, Ramharter M, Djimde AA, Tekete M, Duparc S, Borghini-Fuhrer I, Shin JS, Fleckenstein L. Population Pharmacokinetics of Pyronaridine in Pediatric Malaria Patients. Antimicrob Agents Chemother. 2015 Dec 14;60(3):1450-8. doi: 10.1128/AAC.02004-15. PMID 26666916
- [Derived] Duparc S, Borghini-Fuhrer I, Craft CJ, Arbe-Barnes S, Miller RM, Shin CS, Fleckenstein L. Safety and efficacy of pyronaridine-artesunate in uncomplicated acute malaria: an integrated analysis of individual patient data from six randomized clinical trials. Malar J. 2013 Feb 21;12:70. doi: 10.1186/1475-2875-12-70. PMID 23433102

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PA Group | AL Group
Started | 355 | 180
Completed | 274 | 142
Not Completed | 81 | 38
Not completed — Adverse Event | 6 | 3
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lost to Follow-up | 6 | 1
Not completed — Parasite reappearance/malaria | 67 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PA Group | AL Group | Total
Number analyzed (Participants) | 355 | 180 | 535
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.9 (2.47) | 5.3 (2.52) | 5.0 (2.49)
Age, Customized [Count of Participants; unit: Participants]
  <1 year | 12 | 3 | 15
  1-<5 years | 148 | 69 | 217
  5-12 years | 195 | 108 | 303
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 178 | 96 | 274
  Male | 177 | 84 | 261
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 342 | 172 | 514
  Asian/Oriental | 13 | 8 | 21
Region of Enrollment [Number; unit: participants]
  Gabon | 53 | 27 | 80
  Burkina Faso | 19 | 9 | 28
  Mali | 86 | 44 | 130
  Philippines | 13 | 7 | 20
  Congo, The Democratic Republic of the | 56 | 28 | 84
  Côte D'Ivoire | 72 | 35 | 107
  Kenya | 56 | 30 | 86

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With PCR-Corrected ACPR on Day 28
Description: Percentage of patients with PCR-corrected adequate clinical and parasitological response (ACPR) on Day 28. The PCR-corrected ACPR on Day 28 is defined as the absence of parasitaemia on Day 28 without the patient's meeting any of the criteria of early treatment failure, late clinical failure, or late parasitological failure
Time Frame: Day 28
Population: Efficacy evaluable population: patients who completed a full course of study medication and had a known primary efficacy endpoint at D28; did not miss a dose; did not use concomitant medication, except acetaminophen; did not have a concomitant disease which may interfere with the clear classification of the treatment outcome; did not have a major protocol deviation.C
Measure: Number (95% Confidence Interval); unit: percentage of cured subjects
Arm/Group | PA Group | AL Group
Number analyzed (Participants) | 337 | 167
percentage of cured subjects | 97.6 [95.4 to 99.0] | 98.8 [95.7 to 99.9]
Statistical Analysis 1: Comparison: PA Group; Test type: Other — Analysis of the PCR-corrected ACPR response rate on Day 28 for the PA group. Null hypothesis: The PCR-corrected ACPR response rate on Day 28 for the PA group is ≤90%. Was tested versus the alternative: Alternative hypothesis: The PCR-corrected ACPR response rate on Day 28 for the PA group is >90%; p < 0.0001, Exact binomial test — The threshold for significance was ≤0.025
Statistical Analysis 2: Comparison: PA Group vs AL Group; Null hypothesis: The PCR-corrected ACPR response rate on Day 28 for the PA group is inferior to the PCR-corrected ACPR response rate for the AL group. Was tested versus the alternative: Alternative hypothesis: The PCR-corrected ACPR response rate on Day 28 for the PA group is not inferior to the PCR-corrected ACPR response rate for the AL group; Test type: Non-Inferiority — The secondary efficacy analysis tested the non-inferiority of PA compared to the AL group with regard to the PCR-corrected ACPR response rate on Day 28 using a 2-sided 95% confidence interval (Newcombe Wilson score method without continuity correction) and a 10% non-inferiority margin for the EE population. Non-inferiority was demonstrated if the lower limit of the 2-sided 95% confidence interval for the difference in 28-day PCR-corrected ACPR was not lower than 10%; p = 0.3728, Chi-squared — If non-inferiority of PA was demonstrated, the p-value associated with a superiority test was calculated based on a 2-sided Chi-Square test. If the calculated p-value was <0.05, then the superiority of PA over AL was statistically demonstrated; ACPR percent difference = -1.2, 95% CI 2-sided [-3.6 to 2.1]

2. Secondary Outcome: Percentage of Participants With PCR-Corrected ACPR on Day 14
Description: Percentage of subjects with PCR-corrected adequate clinical and parasitological response (ACPR) on Day 14. The PCR-corrected ACPR on Day 14 is defined as the absence of parasitaemia on Day 14 without the subject's meeting any of the criteria of early treatment failure, late clinical failure, or late parasitological failure
Time Frame: Day 14
Population: Efficacy evaluable population: patients who completed a full course of study medication and had a known primary efficacy endpoint at D28; did not miss a dose; did not use concomitant medication, except acetaminophen; did not have a concomitant disease which may interfere with the clear classification of the treatment outcome; did not have a major protocol deviation.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | PA Group | AL Group
Number analyzed (Participants) | 337 | 167
percentage of subjects | 100.0 [98.9 to 100.0] | 100.0 [97.8 to 100.0]

3. Secondary Outcome: Crude ACPR (Non-PCR Corrected ACPR) (Crude Cure Rate) on Day 14 and Day 28
Description: Percentage of subjects with adequate clinical and parasitological response (ACPR) on Day 14 and 28, without correction by PCR. Crude ACPR on Day 14 and 28 is defined as the absence of parasitaemia on Day 14 and 28 without the subject's meeting any of the criteria of early treatment failure, late clinical failure, or late parasitological failure
Time Frame: Days 14 and 28
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | PA Group | AL Group
Number analyzed (Participants) | 337 | 167
percentage of subjects
  Percentage of Participants with ACPR at Day 14 | 100 [98.9 to 100.0] | 100 [97.8 to 100.0]
  Percentage of Participants with ACPR at Day 28 | 90.2 [86.5 to 93.2] | 89.2 [83.5 to 93.5]

4. Secondary Outcome: Parasite Clearance Time
Description: Parasite clearance time is defined as the time from first dosing to the time of first blood draw with parasite clearance. Parasite clearance was defined as zero presence of asexual parasites for 2 consecutive negative readings taken between 7 and 25 hours apart
Time Frame: Days 0, 3, 7, 14, 21, 28, 35, and 42 or on any other day if the subject spontaneously returned within the 42-day study period
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | PA Group | AL Group
Number analyzed (Participants) | 337 | 167
hours | 24.1 [24.0 to 24.1] | 24.2 [24.0 to 31.8]

5. Secondary Outcome: Fever Clearance Time
Description: Fever clearance time is defined as the time from first dosing to the first normal reading of temperature for 2 consecutive normal temperature readings taken between 7 and 25 hours apart.
Time Frame: Day 0 and every 8 hours over ≥72 hours following first study drug administration or temperature normalization for ≥2 readings between 7 and 25 hours apart, then at each visit and as clinically indicated (within the 42-day study period)
Population: Efficacy evaluable population*: patients who completed a full course of study medication and had a known primary efficacy endpoint at D28; did not miss a dose; did not use concomitant medication, except acetaminophen; did not have a concomitant disease which may interfere with the clear classification of the treatment outcome; did not have a major protocol deviation.
  *does not include subjects initially included on history of fever.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | PA Group | AL Group
Number analyzed (Participants) | 264 | 126
hours | 8.1 [8.0 to 8.1] | 8.1 [8.0 to 15.8]

6. Secondary Outcome: Proportion of Subjects With Cleared Parasites on Days 1, 2, and 3
Description: as for outcome 4
Time Frame: Days 1, 2, and 3
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | PA Group | AL Group
Number analyzed (Participants) | 337 | 167
percentage of subjects
  Percentage of Participants with parasite clearance at Day 1 (24h after first dose) | 49.9 [44.5 to 55.2] | 43.7 [36.2 to 51.2]
  Percentage of Participants with parasite clearance at Day 2 (48h after first dose) | 95.5 [93.3 to 97.8] | 95.2 [92.0 to 98.4]
  Percentage of Participants with parasite clearance at Day 3 (72h after first dose) | 97.0 [95.2 to 98.8] | 98.8 [97.2 to 100.0]

7. Secondary Outcome: Proportion of Subjects With Fever Cleared on Days 1, 2, and 3
Description: as for outcome 5
Time Frame: Days 1, 2, and 3
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | PA Group | AL Group
Number analyzed (Participants) | 264 | 126
percentage of subjects
  Percentage of Participants with fever clearance at Day 1 (24h after first dose) | 87.1 [83.1 to 91.2] | 81.0 [74.1 to 87.8]
  Percentage of Participants with fever clearance at Day 2 (48h after first dose) | 98.5 [97.0 to 100.0] | 96.8 [93.8 to 99.9]
  Percentage of Participants with fever clearance at Day 3 (48h after first dose) | 99.6 [98.9 to 100.0] | 98.4 [96.2 to 100.0]

8. Secondary Outcome: Number of Subjects With ≥1 Adverse Event
Time Frame: Day 0 to 42. Subjects experiencing AEs at Day 42 were followed for up to 30 days after the end of study or resolution of the event, whichever was earlier
Population: Safety population: all randomized subjects who received any amount of study medication. Subjects were analyzed as treated
Measure: Count of Participants; unit: Participants
Arm/Group | PA Group | AL Group
Number analyzed (Participants) | 355 | 180
Participants
  Nr subj. with ≥1 AE | 285 | 143
  Nr subj. with ≥1 treatment-related AE | 132 | 80
  Nr subj. with ≥1 SAE | 1 | 0
  Nr subj. with ≥1 treatment-related SAE | 0 | 0
  Nr subj. with ≥1 severe or life-threatening AE | 2 | 2
  Nr subj. with ≥1 AE leading to death | 0 | 0
  Nr subj. ≥1 AE leading to drug discontinuation | 6 | 3
  Nr subj. with ≥1 AE leading to study withdrawal | 6 | 3

ADVERSE EVENTS:
Time Frame: Day 0 to 42. Subjects experiencing AEs at Day 42 were followed for up to 30 days after the end of study or resolution of the event, whichever was earlier
Groups:
- PA Group: Oral pyronaridine/artesunate (PA, 60:20mg granules) once a day for 3 consecutive days (Days 0, 1, and 2).
  Posology was based on body weight ranges. Subjects were randomized in a 2:1 ratio to receive either PA or AL.
- AL Group: Oral artemether/lumefantrine (AL, 20:120mg crushed tablets) twice a day for 3 consecutive days (Days 0, 1, and 2).
  Posology was based on body weight ranges. Subjects were randomized in a 2:1 ratio to receive either PA or AL.
Arm/Group | PA Group | AL Group
All-Cause Mortality (participants affected / at risk) | 0/355 | 0/180
Serious Adverse Events (participants affected / at risk) | 1/355 | 0/180
Other Adverse Events (participants affected / at risk) | 285/355 | 143/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PA Group (N=355) | AL Group (N=180)
Malaria (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PA Group (N=355) | AL Group (N=180)
Anaemia (Blood and lymphatic system disorders) | 34 (36) | 14 (14)
Splenomegaly (Blood and lymphatic system disorders) | 8 (8) | 4 (5)
Vomiting (Gastrointestinal disorders) | 25 (27) | 8 (9)
Abdominal pain (Gastrointestinal disorders) | 11 (11) | 8 (8)
Pyrexia (General disorders) | 23 (24) | 8 (8)
Influenza like illness (General disorders) | 19 (19) | 8 (8)
Upper respiratory tract infection (Infections and infestations) | 42 (44) | 19 (19)
Bronchitis (Infections and infestations) | 28 (31) | 10 (10)
Helminthic infection (Infections and infestations) | 11 (11) | 3 (4)
Nasopharyngitis (Infections and infestations) | 9 (10) | 3 (3)
Rhinitis (Infections and infestations) | 8 (10) | 3 (3)
Tinea capitis (Infections and infestations) | 7 (7) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4) | 5 (5)
Tonsillitis (Infections and infestations) | 2 (2) | 4 (4)
Platelet count increased (Investigations) | 33 (33) | 19 (19)
Blood glucose decreased (Investigations) | 32 (32) | 19 (19)
Blood albumin decreased (Investigations) | 21 (21) | 16 (16)
Aspartate aminotransferase increased (Investigations) | 17 (17) | 8 (8)
Blood potassium increased (Investigations) | 16 (16) | 6 (6)
Haematocrit decreased (Investigations) | 16 (16) | 5 (5)
Haemoglobin decreased (Investigations) | 15 (15) | 5 (5)
White blood cell count increased (Investigations) | 9 (9) | 2 (2)
Alanine aminotransferase increased (Investigations) | 7 (7) | 2 (2)
Blood creatinine decreased (Investigations) | 7 (7) | 7 (7)
Platelet count decreased (Investigations) | 7 (7) | 1 (1)
Headache (Nervous system disorders) | 13 (14) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 44 (48) | 28 (30)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No